CLINICAL TRIAL: NCT05282862
Title: Guided Surgery for Horizontal Bone Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: ITI Foundation (Industry)
Responsible Party: Principal Investigator, Mihai Tarce, Researcher, PhD student, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S61322
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Edentulous Alveolar Ridge Atrophy
Keywords: implant; bone augmentation; GBR

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freehand (Active Comparator): Conventional bone augmentation using a particulate graft material (DBBM) and a collagen barrier membrane.
  Interventions: Procedure: Horizontal bone augmentation
- Guided (Experimental): Bone augmentation performed using the materials as in the Freehand group, but using a surgical guide to help define the shape of the guide.
  Interventions: Procedure: Horizontal bone augmentation

INTERVENTIONS:
Procedure: Horizontal bone augmentation — Horizontal bone augmentation of a limited span (1-2 teeth) edentulous ridge with neighboring teeth present.

SUMMARY:
The aim of the research project is to develop a novel protocol for guided bone regeneration (GBR) and assess whether such a patient specific 3D printed guide can improve the accuracy of the resulting bone augmentation when compared to conventional freehand protocols.

This study will be an open, prospective, randomized controlled clinical trial. A total of 28 healthy adult patients requiring bone augmentation of an edentulous site with adjacent teeth prior to implant placement will be included in a clinical trial.

All patients have to fulfill all inclusion criteria and none of the exclusion criteria. The total study duration for the patient will be around 7 months, from inclusion to final follow-up.

A virtual plan representing the ideal shape of the augmentation will be prepared. Bone augmentation guides (molds) will be designed and 3D printed for each case. These molds will encompass the defect and the desired augmentation (including the overfill compensating for the expected resorption) on the buccal aspect, leaving a small access space on the coronal aspect of the defect which will be used to insert the grafting material. Additionally, they will have holes near the mesial, distal and apical edges allowing for fixation of the barrier membrane using pin placement when the mold is in position. Finally, they will extend to the occlusal surface of teeth adjacent to the defect site in order to allow precise positioning and will have a protrusion (handle) on the buccal aspect allowing for easier handling and positioning.

The trial will have two groups, a freehand group where conventional bone augmentation surgery will be performed and the clinician will determine the shape of the graft manually, and a guided group where the guide described above will be used. A 50:50 mixture of DBBM and autogenous bone will be used for both groups, resulting in a composite graft. The graft will be covered by a resorbable collagen membrane.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least one site requiring bone augmentation prior to or simultaneously with implant placement;
* the above mentioned site should have adjacent teeth both mesially and distally;
* a history of edentulism in the area of implant treatment of at least 3 months;
* provision of informed consent.

Exclusion Criteria:

* unlikely to be able to comply with the study procedures, as judged by the investigator;
* untreated periodontal disease;
* known or suspected current malignancy;
* history of chemotherapy within 5 years prior to study;
* history of radiation in the head and neck region;
* history of other metabolic bone diseases;
* a medical history that makes bone augmentation or implant insertion unfavorable;
* need for systemic corticosteroids;
* current or previous use of intravenous bisphosphonates;
* current or previous use of oral bisphosphonates;
* history of bone grafting and/or sinus lift in the planned implant area;
* present alcohol and/or drug abuse;
* involvement in the planning and conduct of the study;
* previous enrolment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of resulting graft, immediately post-operatively. | Immediately after surgery
  Linear and volumetric difference between plan and resulting graft, measured on the post-op CBCT.
Accuracy of resulting graft, 6 months after surgery | Six months after surgery
  Linear and volumetric difference between plan and resulting graft, measured on the CBCT taken 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Tarce, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven Sint Rafaël Campus, Leuven, Belgium